CLINICAL TRIAL: NCT03538145
Title: Psychometric Evaluation of the Traditional Chinese Version of Resilience Scale-14 and the Assessment of the Resilience Level of Hong Kong Adolescents
Brief Title: Psychometric Evaluation of the Traditional Chinese Version of Resilience Scale-14
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: UW17-378
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Resilience of Hong Kong Adolescents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will aim to translate the original RS-14 (English version) into traditional Chinese. It will then test the psychometric properties of the newly translated RS-14 to examine its factorial structure using both exploratory factor analysis (EFA) and CFA.

DETAILED DESCRIPTION:
Mental health problems in adolescents reflect a global problem that is becoming more prevalent in Hong Kong. In Hong Kong, there is a significant change in family structure to small nuclear families. Children receive more attention and may even be overprotected by parents. Also, parents' great expectations for high academic achievement also contribute to the increase in mental health problems among adolescents in Hong Kong. The Polytechnic University and the Christian Family Service Centre conducted a mental health survey study of 12,518 Form 1 to Form 7 pupils from 2011 to 2014. Of the respondents, 62.1% demonstrated slight to very serious depression symptoms. Evidence has shown that depressive symptoms predict suicidal tendencies among adolescents.

Resilience effectively prevents the development of mental health problems and is associated with positive mental health outcomes in adolescents. Assessing resilience in adolescents is therefore crucial for developing a thorough understanding of their responses to stress and adversity. The literature reports various instruments used to assess resilience, such as the Connor-Davidson Resilience Scale (CD-RISC) and the Resilience Scale (RS). And translated version of RS-14 is also developed because of linguistic and cultural differences.

The proposed study will aim to translate the original RS-14 (English version) into traditional Chinese. It will then test the psychometric properties of the newly translated RS-14 to examine its factorial structure using both exploratory factor analysis (EFA) and CFA. Furthermore, using the newly validated RS-14, a survey will be conducted to assess the resilience level of a large sample group of Hong Kong Chinese adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Form 1 students (Grade 7, 12 to 13 years of age) from six secondary schools

Exclusion Criteria:

* Those with chronic illnesses or identified cognitive or learning problems will be excluded.

Ages: 12 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Form 1 students (Grade 7, 12 to 13 years of age) from six secondary schools across three major districts (Hong Kong Island, Kowloon and the New Territories) will be randomly selected and invited to participate in the proposed study.
Sampling Method: Non-Probability Sample
Enrollment: 2900 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Resilience level | Baseline
  The RS-14 is a 14-item scale measuring two factors: personal competence, and acceptance of self and life. The item is answered using a 7-point Likert scale ranging from "strongly disagree" to "strongly agree," with total possible scores ranging from 14 to 98. Higher scores indicate higher levels of resilience.

SECONDARY OUTCOMES:
Number of depressive symptoms | Baseline
  The subjects' depressive symptoms will be assessed using the Chinese version of the CES-DC. The CES-DC comprises 20 fully standardized items to evaluate depressive symptoms. All items are evaluated on a four-point self-report scale in relation to their incidence during the last week, which were scored from 0 to 3, with total possible scores ranging from 0 to 60, with higher scores indicating greater symptomatology.
Levels of self-esteem | Baseline
  The subjects' self-esteem will be assessed using the Chinese version of the RSES. The RSES is designed to measure the global self-esteem of children and adolescents. The scale comprises 10 items, rated using a 4-point Likert scale ranging from 1 to 4, with total possible scores ranging from 10 to 40. Higher scores indicate higher levels of self-esteem.

CONTACTS AND LOCATIONS:
Overall Officials: Oi Kwan Joyce Chung, Dr, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chung JOK, Lam KKW, Ho KY, Cheung AT, Ho LK, Xei VW, Gibson F, Li WHC. Psychometric evaluation of the traditional Chinese version of the resilience Scale-14 and assessment of resilience in Hong Kong adolescents. Health Qual Life Outcomes. 2020 Feb 19;18(1):33. doi: 10.1186/s12955-020-01285-4. PMID 32075647